CLINICAL TRIAL: NCT00213213
Title: Effectiveness of Sucrose Analgesia in Reducing Pain Responses in Infants Born to Diabetic and Non-diabetic Mothers: A Randomized Controlled Trial
Brief Title: Using Sugar Water to Relieve Pain in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Anna Taddio/Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000002771; CIHR MCT-63143; ISRCTN23411530
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2005-09

CONDITIONS: Pain; Infant, Newborn; Diabetes
Keywords: sucrose; analgesia; pain; neonates; diabetes
MeSH Terms: conditions — Pain; Diabetes Mellitus; Agnosia | interventions — Sucrose

INTERVENTIONS:
Drug: Sucrose

SUMMARY:
This study will examine the safety and effectiveness of sugar water to relieve pain in newborn infants during painful blood tests and injections. Infants of diabetic mothers who receive repeated blood tests will be compared to infants of healthy mothers who receive routine painful procedures.

We believe that administration of sucrose analgesia for every painful cutaneous procedure performed after delivery will result in less pain during the newborn infant screening test.

ELIGIBILITY:
Inclusion Criteria:

* healthy newborn infants ≥36 weeks gestation
* infants born to mothers with diabetes (type 1, type 2, or gestational diabetes that is diet-controlled or insulin-dependent)and infants born to mothers without diabetes

Exclusion Criteria:

* Admission to the neonatal intensive care unit
* plan to undergo circumcision during the study period
* major congenital or neurological anomalies
* clinical diagnosis of birth asphyxia or seizures
* receiving analgesics or sedatives

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240
Dates: Start 2003-07; Study Completion 2005-07

PRIMARY OUTCOMES:
- Infant pain score during the newborn screening test, assessed by the Premature Infant Pain Profile (PIPP), or individual parameters of PIPP (facial grimace, heart rate, oxygen saturation)

SECONDARY OUTCOMES:
(effectiveness):
- Effectiveness of sucrose for repeated heel lances
- Effectiveness of sucrose in decreasing anticipatory pain responses during venipuncture
- Effectiveness of sucrose in decreasing pain response during Vitamin K injection
- Determination of relationship between painful procedures and infant response during routine care procedures
(safety):
- Incidence of vomiting during administration of sucrose
- Oxygen saturation during administration of sucrose
- Serum Glucose concentrations in infants of diabetic mothers

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Taddio A, Shah V, Hancock R, Smith RW, Stephens D, Atenafu E, Beyene J, Koren G, Stevens B, Katz J. Effectiveness of sucrose analgesia in newborns undergoing painful medical procedures. CMAJ. 2008 Jul 1;179(1):37-43. doi: 10.1503/cmaj.071734. PMID 18591525